CLINICAL TRIAL: NCT01898507
Title: Nicotine Metabolism and Low Nicotine Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Andrew Strasser, Research associate professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 816228
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Smoking
Keywords: low nicotine; cigarettes; NMR
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Masking Description: All subjects were blinded to the nicotine content of the study cigarettes.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low nicotine cigarettes (Experimental): Participants will smoke their own brand cigarettes during a baseline 5 day period, followed by a 15-day period of smoking low nicotine content cigarette level 1: 0.25 mg nicotine content, followed by a 15-day period of smoking low nicotine content cigarette level 2: 0.08 mg nicotine content.
  Other: Low nicotine cigarettes
  Interventions: Other: Low nicotine cigarettes

INTERVENTIONS:
Other: Low nicotine cigarettes — 15-day period of smoking low nicotine content cigarette level 1: 0.25 mg nicotine content, followed by a 15-day period of smoking low nicotine content cigarette level 2: 0.08 mg nicotine content.

SUMMARY:
This study examines the effects of smoking low nicotine cigarettes in different groups of smokers. The investigators are focusing on differences in how smokers' bodies break down and eliminate nicotine from their systems. Some people are fast metabolizers of nicotine, meaning they break down and eliminate nicotine from their bodies more quickly. Other people are slower metabolizers meaning they break down and eliminate nicotine more slowly. The investigators are comparing these two groups of smokers for their responses to low nicotine cigarettes. The investigators hypothesize that individuals who smoke low nicotine cigarettes may smoke more intensely or smoke more each day, thereby maintaining their desired nicotine levels, and as a result continue to be exposed to significant toxin levels.

DETAILED DESCRIPTION:
This study examines the effects of smoking low nicotine cigarettes on smoking behaviors and toxin exposure in fast and slow nicotine metabolizing smokers. We will recruit current smokers (split between slow and rapid nicotine metabolizing smokers) for a 35-day protocol. Participants will smoke their own brand cigarettes during a baseline 5 day period, followed by a 15-day period of smoking low nicotine content cigarette level 1: 0.25 mg nicotine content, followed by a 15-day period of smoking low nicotine content cigarette level 2: 0.08 mg nicotine content. This application is designed to provide empirical science to inform the FDA on the effect smoking low nicotine content cigarettes will have on use patterns and harm exposure.

ELIGIBILITY:
Inclusion Criteria:

1. adults age 21-65.
2. smoking at least 10 cigarettes per day.
3. smoking daily for the last 5 years.
4. Provide a baseline breath CO reading equal to or greater than 10 parts per million.
5. smoke predominantly non-menthol filtered cigarettes (research cigarettes are only non-menthol).
6. not currently using any other nicotine containing products such as cigars, smokeless tobacco, nicotine replacement therapies (patch or gum).
7. are fluent in English and are capable of providing written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Participants who meet the inclusion/exclusion criteria and attend an Intake Visit for medical screening will be asked to provide a blood sample to determine NMR. Only those individuals who are characterized as slow or rapid, based on NMRs ≤ .26, or ≥ .42, will be eligible.

Exclusion Criteria:

1. use of any nicotine containing products other than cigarettes
2. current or impending enrollment in smoking cessation program
3. history in the last year or current treatment of substance abuse (other than nicotine dependence)
4. positive drug screen for cocaine, methamphetamines or opiates for urine drug screen at intake session
5. alcohol use greater than 25 standard drinks per week
6. current or planned pregnancy or lactating
7. history or current diagnosis of psychosis, bipolar disorder, mania, or schizophrenia
8. current major depression (history of major depression but in remission for a minimum 6 months is eligible).
9. serious or unstable disease within past year (e.g. cancer other than melanoma, heart disease)
10. history or current diagnosis of COPD
11. history of stroke or heart attack
12. age less than 21 years- We wish to recruit smokers with well established smoking patterns and will restrict recruitment to those over 21
13. age more than 65 years - smoking is often associated with cardiovascular and pulmonary obstructive diseases that manifest later in life. As smokers develop these problems, smoking behavior and biomarkers of harm may be affected therefore we will restrict enrollment to those under age 65
14. provide baseline CO reading less than 10 at initial session
15. current use (or use within past 14 days) of any medication that affects the biotransformation of nicotine, such as anticonvulsant drugs, rifampin, and disulfiram; or any psychoactive medications which can affect smoking behaviors
16. any conditions viewed by the PI or study physician as creating a potential increased risk to a participant due to their participation will be reasons for exclusion
17. at the discretion of the PI, any participants viewed as non-compliant will be excluded from further participation
18. Smoke cigarettes with a filter size other than standard or slim sized as the topography mouthpieces are sized for standard filters and have an adapter for slim cigarettes only.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Smoking topography- total puff volume | up to 35 days

SECONDARY OUTCOMES:
Daily cigarette consumption | Study day 0, 5, 10, 15, 20, 25, 30, 35
  Total number of cigarettes smoked each day.
Urine nicotine metabolite measures | Assessed at Days 5, 20 and 35
  NNK, mercapturic acid metabolites, total nicotine equivalents
Carbon monoxide measurements | Study day 0, 5, 10, 15, 20, 25, 30, 35

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States